CLINICAL TRIAL: NCT04797091
Title: Kidney in Coronavirus Disease 2019 Registry
Acronym: KidneyCOVID19
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Principal Investigator, University of Cologne
Other Study IDs: Kidney in COVID-19
Record Dates: First submitted 2020-04-16; First posted 2021-03-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Corona Virus Infection; SARS-CoV 2
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with SARS-CoV-2-infection: Patients with evidence of SARS-CoV-2-infection
  Interventions: Other: Retrospective data collection
- Control group: Controls will be identified retrospectively at the same hospitals that based on matching of demographics, underlying diseases and duration of hospitalization.
  Interventions: Other: Retrospective data collection

INTERVENTIONS:
Other: Retrospective data collection — Retrospective data collection to overcome the lack of knowledge on epidemiology, clinical course including diagnostic and therapeutic approaches and prognostic factors for SARS-CoV-2-infections and their complications among nephrology and elderly patients, as well as to serve as a platform for future studies and outbreak situations.

SUMMARY:
The SARS-CoV-2 virus is a virus newly identified in January 2020. The WHO defined COVID-19 as a health emergency of international importance. The clinical manifestation of the COVID-19 disease cannot be fully described in the short time.

First insights in patients suffering from acute kidney injury (AKI) during COVID-19 indicate severe course with high mortality. The locally varying spread of SARS CoV-2 infection requires a better understanding of clinical course of COVID-19 in order to be able to establish future treatment approaches.

The examination of attributable mortality and costs of COVID-19 will need to be studied on a multinational basis and therefore Kidney in COVID-19 Registry will particularly use a matched case control design.

DETAILED DESCRIPTION:
The SARS-CoV-2 virus is a virus newly identified in January 2020 in Wuhan, China, which belongs to the group of coronaviruses and causes COVID-19. Due to the rapid spread worldwide, high morbidity and virulence the of causing SARS-CoV-2 , the WHO defined COVID-19 as a health emergency of international importance in February 2020. Due to the rapid spread of the new virus, a comprehensive understanding of the transmission, the course of the disease, the diagnosis and the therapeutic regimen is of the utmost importance. Initial case reports indicate that human-to-human transmission takes place through droplet infection. In contrast to previously known infections from the group of coronaviruses, the SARS-CoV-2 virus has a high ability to infect with already mild symptoms resulting in frequent outbreak situation of worldwide importance. Furthermore, high viral loads are found in the upper respiratory tract of infected people leading to the high virulence of causing SARS-CoV-2. The clinical manifestation of the COVID-19 disease cannot be fully described in the short time. However, symptoms of SARS-CoV-2 virus infection are described with mild symptoms like fever, muscle pain, and dry cough as well as severe complications like virus pneumonia, Acute Respiratory Distress Syndrome (ARDS) and death. Interestingly older and chronically ill patients in particular have a severe course of COVID-19 with intensive care treatment and high mortality. At present, there is no specific therapy available for COVID-19. Treatment approaches are primarily supportive with admission of patients to the intensive care unit (ICU), mechanical ventilation, extracorporeal membrane oxygenation (ECMO) and maintenance of fluid and electrolyte balance. Patients with severe renal insufficiency and fluid retention, pulmonary edema or hyperkalemia may require dialysis. First insights in patients suffering from acute kidney injury (AKI) during COVID-19 indicate severe course with high mortality. First case reports do not describe a beneficial effect of antiviral therapy. The locally varying spread of SARS CoV-2 infection requires a better understanding of clinical course of COVID-19 in order to be able to establish future treatment approaches. Investigators have to attach great importance to high-risk cohorts like patients suffering from chronic renal disease with many comorbidities or patients after kidney transplantation under immunosuppressive drug treatment. Although COVID-19 has been studied for only a few month it is known that especially these patients develop a severe clinical course. Due to increasingly frequent outbreak situations and globally chances in species distributions, local, as well as worldwide surveillances in epidemiology and species distribution are urgently needed. As the clinical course of COVID-19 disease is dependent on the causing viral pathogen and the full picture of clinical manifestation is not yet understand further studies with regard to the disease course are mandatory.

Additionally, the examination of attributable mortality and costs of COVID-19 will need to be studied on a multinational basis and therefore Kidney in COVID-19 Registry will particularly use a matched case control design.

ELIGIBILITY:
Inclusion Criteria:

* Virology evidence of SARS-CoV-2-infection
* Pathological evidence of SARS-CoV-2-infection

Exclusion Criteria:

* Occurrence of ARDS (acute respiratory distress syndrome) without evidence of SARS-CoV-2 infection
* Acute kidney injury without evidence of SARS-CoV-2 infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Particularly, controls will be identified retrospectively at the same hospitals that based on matching of demographics, underlying diseases and duration of hospitalization (i.e. one control per case, both in the same hospital).
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Determination of the global incidence of SARS-CoV-2 infections | 6 months
  Determination of the global incidence of SARS-CoV-2 infections and the resulting effects on kidney function as well as monitoring of global and local developments over time.

SECONDARY OUTCOMES:
Determination of the incidence of acute kidney damage in the context of SARS-CoV2 infections | 6 months
  Determination of the incidence of acute kidney damage in the context of SARS-CoV2 infections
Identification of risk groups and risk factors | 6 months
  Identification of risk groups and risk factors by examining SARS-CoV-2 infections in patients with chronic kidney disease and kidney transplantation
Documentation of mortality rates due to SARS-CoV-2 infections | 6 months
  Documentation of mortality rates in % in comparison to case controls enrolled in the same hospital
Documentation of additional costs due to SARS-CoV-2 infections | 6 months
  Documentation of additional costs in euros in comparison to case controls enrolled in the same hospital
To assess increasing costs associated with SARS-CoV-2-infections | 6 months
  To assess increasing costs associated with SARS-CoV-2-infections
To analyze the effect of SARS-CoV-2-infections on the kidney by means of eGFR | 6 months
  To analyze the effect of SARS-CoV-2 infections on kidney function as determined by estimated Glomerular Filtration Rate (eGFR) after SARS-CoV-2 infection
To analyze the effect of SARS-CoV-2-infections on the kidney by means of maximum creatinine | 6 months
  To analyze the effect of SARS-CoV-2 infections on kidney function as determined by maximum creatinine after SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, PD MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No